CLINICAL TRIAL: NCT07366268
Title: Clinical Evaluation of Topical Apremilast Nanoparticles in the Treatment of Plaque Psoriasis: Clinical, Histopathological and Immunohistochemical Study
Brief Title: Evaluation the Topical Apremilast Nanoformulation in Treatment of Localized Plaque Psoriasis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aliaa Effat Saied Sayed, Assistant lecturer, Assiut University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Nano Apremilast in psoriasis
Record Dates: First submitted 2026-01-10; First posted 2026-01-26 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Psoriasis
Keywords: Psoriasis; Apremilast; Nanotechnology; Topical
MeSH Terms: conditions — Psoriasis | interventions — Betamethasone Valerate

STUDY DESIGN:
Intervention Model Description: Each Participant will receive the different treatment included within the study( intrapatient study)
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Topical Apremilast Nanoformula (Experimental): Participants will receive topical apremilast nanoformula 0.3% applied twice daily for 12 weeks.
  Interventions: Drug: Apremilast Nanoformula 0.3٪
- Topical betamethasone valerate (Active Comparator): Participants will receive topical betamethasone valerate 0.1% cream applied twice daily for 12 weeks.
  Interventions: Drug: betamethasone valerate 0.1% cream
- Combination therapy (Experimental): Participants will receive combined topical apremilast nanoformula 0.3% and topical betamethasone valerate 0.1% cream applied for 12 weeks.
  Interventions: Drug: Apremilast Nanoformula 0.3٪; Drug: betamethasone valerate 0.1% cream

INTERVENTIONS:
Drug: Apremilast Nanoformula 0.3٪ — the nano based formula of apremilast will be prepared from its raw powder at Assuit international center of nanomedicine, Alrajhy Liver hospital, Assuit university. Nanoparticles loaded-apremilast 0.3% will be filled into sealed containers labeled as (number 1) and provided to patients and they will be instructed to apply thin a film twice daily for 12 weeks
  Arms: Combination therapy; Topical Apremilast Nanoformula
Drug: betamethasone valerate 0.1% cream — • Betamethsone valerate cream 0.1%: The commercially available betamethasone valerate cream will be re-packaged into identical, non-identifiable containers labeled (number 2 ) in order to ensure patient blinding and it will be applied twice daily for 12 weeks
  Arms: Combination therapy; Topical betamethasone valerate

SUMMARY:
This study is a comparative randomized clinical trial evaluating the efficacy and safety of topical apremilast nanoemulsion 0.3% in the treatment of localized mild to moderate plaque psoriasis.Clinical efficacy will be assessed using TES score, Physician Global Assessment (PGA), dermoscopy, and patient satisfaction, while safety is monitored through adverse effect reporting. In addition, histopathological and immunohistochemical evaluation of PDE4 expression will be performed before and after treatment to assess tissue-level responses.

The study aims to determine whether topical apremilast nano-formulation, alone or combined with corticosteroids, offers an effective and safer alternative to conventional topical therapy, with improved local efficacy and reduced corticosteroid-related adverse effects.

DETAILED DESCRIPTION:
Psoriasis is a chronic immune-mediated inflammatory skin condition with a strong genetic predisposition and an autoimmune pathogenic characteristic . Its worldwide prevalence is up to 2% but this varies between different geographic regions . In Egypt, the prevalence of psoriasis ranges between 0.19% and 3% .

Individuals with psoriasis frequently endure marked psychological distress. This includes social embarrassment, reduced self esteem, anxiety, depression, and an increased tendency toward suicidal ideation and behavior .

Psoriasis Skin lesions are usually symmetrical, sharply demarcated, with red or pink raised plaques, and covered with silvery scales. These plaques reflect key pathological processes, including inflammation, keratinocyte hyperproliferation, and angiogenesis .

Cellular responses to environmental stimuli and intracellular signaling in various cell types-including myeloid, lymphoid, and other inflammatory cells-are mediated by intracellular "second messengers," particularly cyclic adenosine monophosphate (cAMP) .

Phosphodiesterase4 (PDE4) is one of the major cAMP-selective PDEs expressed in epithelial cells . It is also present in several mesenchymal cell types, including dermal keratinocytes, smooth muscle cells, vascular endothelial cells, and chondrocytes, By decreasing intracellular cAMP, PDE4 promotes production of pro-inflammatory mediators and decreases production of anti-inflammatory mediators. Conversely, inhibition of PDE4 increases the intracellular concentration of cAMP and selectively blocks pro-inflammatory cytokines, such as TNF-α, IFN-γ, and IL-2 production from peripheral blood monocytes and T cells.

PDE4 has four subtypes (A, B, C and D). These subtypes are encoded on separate genes. Expression of the PDE4A subtype increased in nearly all cell types of the skin of psoriasis patients. PDE4B is present in vessels and in immune cells, whereas PDE4D is expressed in fibroblasts and endothelial cells .

Management of mild to moderate psoriasis usually begins with topical therapies, including emollients, topical corticosteroids, calcipotriol, tar preparations, and dithranol. There is little evidence to guide the selection of topical treatments, so it can be based on patient and prescriber preference .

Topical glucocorticoids are the first-line therapy in mild to moderate psoriasis and areas where other topical treatments may cause irritation, such as joints or genitals . Corticosteroids bind to intracellular corticosteroid receptor and regulate gene transcription of numerous genes, particularly those that code for pro-inflammatory cytokines. They act as vasoconstrictive, antiproliferative, anti-inflammatory and immunosuppressive.

However, long-term application of topical corticosteroids may cause skin atrophy, striae, telangiectasia, adrenal suppression and hypopigmentation. Additionally, abrupt discontinuation can precipitate early disease relapse or rebound flares.

Apremilast is classified as a small-molecule phosphodiesterase4 (PDE4) inhibitor , It inhibits PDE4 isoforms from all four sub-families (A,B,C,D) Apremilast acts by hindering the conversion of cyclic adenosine monophosphate (cAMP) to AMP . further causing an intracellular accumulation of cyclic adenosine monophosphate (cAMP) causing a reduction in the production of inflammatory mediators such as CX-CL9, CX-CL10, IFN-γ, TNF-α, IL-2, IL-8, IL-12, and IL-23, thereby attenuating the inflammatory cascade .

Its oral form is FDA approved for plaque psoriasis in adult patients eligible for systemic therapy or phototherapy, as well as for adults with moderately to severely active psoriatic arthritis. . It is recommended that apremilast be titrated to the recommended dose of 30 mg twice daily, to be taken orally starting on day 6 .

The results of long-term, placebo-controlled study (ESTEEM 2) established the efficacy of oral apremilast in patients with plaque psoriasis, and are consistent with those reported in ESTEEM 1.The primary end point in this study was met, with a significantly greater proportion of patients treated with apremilast achieving a PASI 75 response at week 16 vs. placebo. Across different phases of study, PASI 75 responses at week 16 have ranged from 29% to 41%.

Apremilast is low soluble and low permeable classifying the drug as biopharmaceutical classification system (BCS) class 4 molecule with a poor solubility of 10-14 μg/mL. The oral medication of apremilast has systemic side effects such as diarrhea, nausea, vomiting, weight loss, and depression in some cases .

These limitations highlight the need for alternative routes of administration that enhance drug delivery to affected skin while minimizing systemic exposure. Topical delivery of apremilast represents a promising strategy to achieve localized therapeutic effects with fewer systemic side effects and improve patient outcomes .

Nevertheless, poor solubility and limited skin penetration restrict the effectiveness of topical apremilast, particularly in psoriatic skin, which is thickened and inflamed . Hence, the incorporation into nanotechnology-based drug delivery systems could be used as a strategy to improve its solubility and permeability in order to improve dermal bioavailability and consequently to achieve local anti-inflammatory efficacy .

Several ex vivo studies have demonstrated that apremilast loaded nanoparticles significantly increase skin retention compared with conventional gel formulations, resulting in improved therapeutic outcomes. Cytotoxicity and skin irritation studies further indicate that nano formulations are safe and well tolerated .

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥18 years.
* Pattern: Patients with chronic plaque psoriasis not exceeding 10% of the body surface area.

Exclusion Criteria:

* History of phototherapy or systemic treatment in the previous 12 weeks, topical psoriasis treatment within the last 4 weeks.
* Renal, hepatic disease, cardiovascular, Immunosuppressive therapy, endocrine and blood disease or mental illness.
* Pregnancy, breast-feeding or women planning to become pregnant within 3 months.
* Psoriasis exceeding 10% of body surface area or other severe types of psoriasis requiring systemic treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Change in Psoriasis thickness,erythema, and scaling (TES score) from baseline to Week 12 | Baseline to week 12 and two months after to detect recurrence .
  To evaluate the efficacy and safety of topical apremilast nanoemulsion 0.3٪ for treatment of localized plaque psoriasis as a monotherapy versus topical betamethasone valerate 0.1٪ cream alone and its combination with a topical betamethasone valerate 0.1٪ cream

SECONDARY OUTCOMES:
Change in dermoscopic features of psoriatic plaques from baseline to Week 12 | Baseline to week 12
Change in histopathological features of psoriatic plaques from baseline to Week 12 | Baseline to week 12
Change in immunohistochemical expression of PDE4( B/C/D) from baseline to Week 12 | Baseline to week 12

REFERENCES:
- [Background] Delestras S, Roustit M, Bedouch P, Minoves M, Dobremez V, Mazet R, Lehmann A, Baudrant M, Allenet B. Comparison between two generic questionnaires to assess satisfaction with medication in chronic diseases. PLoS One. 2013;8(2):e56247. doi: 10.1371/journal.pone.0056247. Epub 2013 Feb 20. PMID 23437104
- [Background] Nestor MS, Fischer D, Arnold D. Randomized, Investigator-Blinded Study to Compare the Efficacy and Tolerance of a 650-microsecond, 1064-nm YAG Laser to a 308-nm Excimer Laser for the Treatment of Mild to Moderate Psoriasis Vulgaris. J Drugs Dermatol. 2020 Feb 1;19(2):176-183. doi: 10.36849/JDD.2020.4769. PMID 32129962
- [Background] Louden BA, Pearce DJ, Lang W, Feldman SR. A Simplified Psoriasis Area Severity Index (SPASI) for rating psoriasis severity in clinic patients. Dermatol Online J. 2004 Oct 15;10(2):7. PMID 15530297
- [Background] Parmar PK, Bansal AK. Novel nanocrystal-based formulations of apremilast for improved topical delivery. Drug Deliv Transl Res. 2021 Jun;11(3):966-983. doi: 10.1007/s13346-020-00809-1. PMID 32588281
- [Background] Rapalli VK, Tomar Y, Sharma S, Roy A, Singhvi G. Apremilast loaded lyotropic liquid crystalline nanoparticles embedded hydrogel for improved permeation and skin retention: An effective approach for psoriasis treatment. Biomed Pharmacother. 2023 Jun;162:114634. doi: 10.1016/j.biopha.2023.114634. Epub 2023 Apr 3. PMID 37018989
- [Background] Sarango-Granda P, Silva-Abreu M, Calpena AC, Halbaut L, Fabrega MJ, Rodriguez-Lagunas MJ, Diaz-Garrido N, Badia J, Espinoza LC. Apremilast Microemulsion as Topical Therapy for Local Inflammation: Design, Characterization and Efficacy Evaluation. Pharmaceuticals (Basel). 2020 Dec 21;13(12):484. doi: 10.3390/ph13120484. PMID 33371334
- [Background] Papp K, Cather JC, Rosoph L, Sofen H, Langley RG, Matheson RT, Hu C, Day RM. Efficacy of apremilast in the treatment of moderate to severe psoriasis: a randomised controlled trial. Lancet. 2012 Aug 25;380(9843):738-46. doi: 10.1016/S0140-6736(12)60642-4. Epub 2012 Jun 29. PMID 22748702
- [Background] Papp K, Reich K, Leonardi CL, Kircik L, Chimenti S, Langley RG, Hu C, Stevens RM, Day RM, Gordon KB, Korman NJ, Griffiths CE. Apremilast, an oral phosphodiesterase 4 (PDE4) inhibitor, in patients with moderate to severe plaque psoriasis: Results of a phase III, randomized, controlled trial (Efficacy and Safety Trial Evaluating the Effects of Apremilast in Psoriasis [ESTEEM] 1). J Am Acad Dermatol. 2015 Jul;73(1):37-49. doi: 10.1016/j.jaad.2015.03.049. PMID 26089047
- [Background] Paul C, Cather J, Gooderham M, Poulin Y, Mrowietz U, Ferrandiz C, Crowley J, Hu C, Stevens RM, Shah K, Day RM, Girolomoni G, Gottlieb AB. Efficacy and safety of apremilast, an oral phosphodiesterase 4 inhibitor, in patients with moderate-to-severe plaque psoriasis over 52 weeks: a phase III, randomized controlled trial (ESTEEM 2). Br J Dermatol. 2015 Dec;173(6):1387-99. doi: 10.1111/bjd.14164. Epub 2015 Nov 7. PMID 26357944
- [Background] Schafer PH, Parton A, Capone L, Cedzik D, Brady H, Evans JF, Man HW, Muller GW, Stirling DI, Chopra R. Apremilast is a selective PDE4 inhibitor with regulatory effects on innate immunity. Cell Signal. 2014 Sep;26(9):2016-29. doi: 10.1016/j.cellsig.2014.05.014. Epub 2014 May 29. PMID 24882690
- [Background] Ahmed SS, Manchanda Y, De A, Das S, Kumar R. Topical Therapy in Psoriasis. Indian J Dermatol. 2023 Jul-Aug;68(4):437-445. doi: 10.4103/ijd.ijd_422_23. PMID 37822388
- [Background] Chan JJ. Psoriasis: an update on topical and systemic therapies. Aust Prescr. 2025 Jun;48(3):87-92. doi: 10.18773/austprescr.2025.026. PMID 40568686
- [Background] Schafer PH, Truzzi F, Parton A, Wu L, Kosek J, Zhang LH, Horan G, Saltari A, Quadri M, Lotti R, Marconi A, Pincelli C. Phosphodiesterase 4 in inflammatory diseases: Effects of apremilast in psoriatic blood and in dermal myofibroblasts through the PDE4/CD271 complex. Cell Signal. 2016 Jul;28(7):753-63. doi: 10.1016/j.cellsig.2016.01.007. Epub 2016 Jan 22. PMID 26806620
- [Background] Ponikowska M, Vellone E, Czapla M, Uchmanowicz I. Challenges Psoriasis and Its Impact on Quality of Life: Challenges in Treatment and Management. Psoriasis (Auckl). 2025 May 1;15:175-183. doi: 10.2147/PTT.S519420. eCollection 2025. PMID 40330837
- [Background] Parisi R, Iskandar IYK, Kontopantelis E, Augustin M, Griffiths CEM, Ashcroft DM; Global Psoriasis Atlas. National, regional, and worldwide epidemiology of psoriasis: systematic analysis and modelling study. BMJ. 2020 May 28;369:m1590. doi: 10.1136/bmj.m1590. PMID 32467098